CLINICAL TRIAL: NCT03209765
Title: Effectiveness of WhatsApp Reminder on Compliance of Colorectal Cancer Screening: a Randomized Controlled Study
Brief Title: WhatsApp Reminder on FIT Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Thomas Yuen Tung Lam, Nursing Officer, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: WhatsApp Compliance Study
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer; Screening Compliance; Fecal Immunochemical Test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp reminder (Active Comparator): An interactive WhatsApp reminder to return to the centre for taking faecal tubes for screening
  Interventions: Other: WhatsApp reminder
- No reminder (No Intervention)

INTERVENTIONS:
Other: WhatsApp reminder — An interactive WhatsApp reminder to return to the centre for taking faecal tubes for screening
  Arms: WhatsApp reminder

SUMMARY:
It is estimated that there are about 1.4 million patients with colorectal cancer (CRC) worldwide, with a rising trend in CRC incidence in many Asian Pacific countries. In Hong Kong, colorectal cancer ranks first in cancer incidence and second in cancer mortality based on data from 2014.

Recent guidelines from USA, Europe and Asia Pacific region recommend CRC screening for average-risk asymptomatic individuals starting at age 50. Fecal immunochemical tests (FIT), is one of the recommendation as first-line modality for CRC screening. Since yearly testing is recommended to maintain programmatic effectiveness longitudinal adherence is a critical component of FOBT-based screening programs. Our previous study conducted in Hong Kong showed that the rate of compliance with CRC screening was declining since the first year of enrolment8.

In recent years, social media (SM) has become an increasingly popular source of health information. By providing an easily accessible and interactive channel of communication between reviewers and information providers, it has potential values for affecting public health. However, the effects of SM on the compliance of CRC screening by FIT has not yet been studied.

WhatsApp Messenger, is the most popular social media messaging app worldwide. This randomized controlled study will investigate the effect of WhatsApp vs no reminder on the compliance of CRC screening by FIT.

DETAILED DESCRIPTION:
It is estimated that there are about 1.4 million patients with colorectal cancer (CRC) worldwide, with a rising trend in CRC incidence in many Asian Pacific countries. In Hong Kong, colorectal cancer ranks first in cancer incidence and second in cancer mortality based on data from 2014.

Recent guidelines from USA, Europe and Asia Pacific region recommend CRC screening for average-risk asymptomatic individuals starting at age 50. Fecal immunochemical tests (FIT), is one of the recommendation as first-line modality for CRC screening. Since yearly testing is recommended to maintain programmatic effectiveness longitudinal adherence is a critical component of FOBT-based screening programs. Our previous study conducted in Hong Kong showed that the rate of compliance with CRC screening was declining since the first year of enrolment8.

In recent years, social media (SM) has become an increasingly popular source of health information. By providing an easily accessible and interactive channel of communication between reviewers and information providers, it has potential values for affecting public health. However, the effects of SM on the compliance of CRC screening by FIT has not yet been studied.

WhatsApp Messenger, is the most popular social media messaging app worldwide. This randomized controlled study will investigate the effect of WhatsApp vs no reminder on the compliance of CRC screening by FIT.

All subjects will be recruited from the existing cohort of screening participants who joined the bowel cancer screening programme in the CUHK JC Bowel Cancer Education Centre in 2016 with FOBT negative in the first round of screening, and who are expected to follow-up and return to the centre in 2017 for their second round of FOBT screening.

Each study subjects will be offered either an interactive WhatsApp reminder to return to the centre for taking faecal tubes for screening; or usual care, where no additional intervention will be offered. A simple random sampling process will be administered using computer-generated numbers so that each participant will have a 50% probability for assignment into each group. All potential participants identified who are eligible for the study will be randomized by a computer randomizer, which will give a number indicating the group assigned.

The outcome of interest included the proportion of subjects who return to the centre and retrieve faecal tubes for screening 30 days within the scheduled time for the second year of the screening test.

To investigate the long-term effect of WhatsApp reminder on FIT compliance, all subjects in this study (except those died or had positive FIT result) will be called in the first quarter of 2019 and offered FIT again in a cross-over design in 2019, i.e. 1) patients initially randomized to WhatsApp reminder group in 2017 will receive no reminder in 2019; and 2) those randomized to no reminder group in 2017 will receive WhatsApp reminder in 2019.. The FIT pickup and return rate and reason of default will be recorded again.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who joined the bowel cancer screening programme in the CUHK JC Bowel Cancer Education Centre and are expected to follow up for annual FIT.

Exclusion Criteria:

* Lack of access to WhatsApp Messenger

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Compliance rate | 1 year
  Compliance rate of FIT in the year of receiving the interventions/control

SECONDARY OUTCOMES:
Compliance rate of second round | 3 years
  Compliance rate of FIT in the year of second round of follow up after crossing over

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yuen Tung Lam, MSc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided